CLINICAL TRIAL: NCT05226195
Title: The Effect of Kinesio® Taping on Post-Surgical Functional Outcomes in Patients Undergoing Total Knee Replacement Surgery
Brief Title: Effect of Kinesio® Taping in Total Knee Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nihan Ozunlu Pekyavas, Associated Proffesor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA21/464
Record Dates: First submitted 2022-01-13; First posted 2022-02-07 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis; Post-Surgical Complication
Keywords: Kinesiotape; Post-Surgical Functional Outcomes; Total Knee Replacement Surgery
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Sterile Kinesio tape application (Experimental): The standard post-surgical protocol and sterile EDF kinesio-taping will be applied to this group. The clinical evaluation will be made on the 15th, 45th and 90th days; functional measurements will be taken. The follow-up period was determined as 3 months.
  Interventions: Other: Sterile Kinesio Taping
- Group 2: Control group (No Intervention): The standard post-surgical protocol applied in our clinic will be applied to Group 2. The clinical evaluation will be made on the 15th, 45th and 90th days; functional measurements will be taken. The follow-up period was determined as 3 months.

INTERVENTIONS:
Other: Sterile Kinesio Taping — The standard post-surgical protocol and sterile EDF kinesio-taping will be applied to this group in the operating room at the end of the surgery in a sterile manner according to the epidermis-dermis-fascia (EDF) technique previously described in the literature (without tension). Original KinesioTex® Tape will be used in the study. The day of taping will be considered as Day 0 and the tapes will be changed on the 4th day, the 7th day.
  Arms: Group 1: Sterile Kinesio tape application

SUMMARY:
Total knee replacement, which is the gold standard surgical treatment method applied in today's conditions, in order to maintain the patient's daily life without pain, to provide the knee joint range of motion, to eliminate the deformity and instability in the knee joint in advanced stage (Stage 3-4) knee osteoarthritis (OA) that does not benefit from conservative treatment. Obtaining the best clinical outcome for the patient after surgery is only possible with the implementation of post-surgical physical therapy and rehabilitation programs.

Edema and pain occurring in the early post-surgical period prevent patients from moving freely, and as a result, the psychological state of the patients is also affected. With effective physiotherapy, besides relieving pain and edema, patients' sensorimotor performances, proprioceptive senses and body balances are restored, and thus the brain is taught how to maintain joint functions. For this reason, new physiotherapy methods are being developed every day for this purpose.

"Kinesio Taping" (KT) is one of the modern physiotherapy methods that has been widely used in sports orthopedics in recent years. It was developed by Kenzo Kase in 1973 and is used clinically to relieve pain and edema, and to increase motor function in musculoskeletal diseases. In this method, an adhesive cotton-based tape called kinesio tape is used. The elastic structure of this band, which allows it to extend 130-140% of its original length, similar to the skin, together with its three-dimensional "fingerprint" texture specific to the band, causes the formation of microfolds on the skin. The formation of these folds; It is known that it increases the proprioceptive perception of the related joint by stimulating skin mechanoreceptors. It also reduces the pressure under the skin and helps relieve pain by increasing lymphatic drainage. The Epidermis-Dermis-Fascia (EDF) taping method is a KB method that has been developed in recent years. It provides less tension and is more easily applied to painful areas. The narrow strips of the applied tape provide more stimulation in the most superficial tissues5. Although studies on the effect of other application methods on rehabilitation after knee replacement surgery are available in the literature, there is no study in the literature showing the effects of the EDF technique.

In this study, it is aimed to evaluate the effect of KT applied with EDF technique on clinical results in the early postoperative period in patients who have undergone total knee replacement surgery. The hypothesis of this study is; It was determined that "pain and edema decrease and functional gain increases in patients who underwent KT after total knee prosthesis surgery".

ELIGIBILITY:
Inclusion Criteria:

* to be volunteered to participate in the study.
* It will be performed in patients who have stage 3-4 osteoarthritis according to the "Kellgren-Lawrence" classification and therefore undergo total knee replacement surgery in a ligament-cutting design in the Department of Orthopedics and Traumatology of Baskent University Ankara Hospital.

Exclusion Criteria:

* Patients who underwent total knee prosthesis surgery in a hinge-preserving and hinged design
* Patients who underwent simultaneous bilateral total knee prosthesis surgery
* Patients with lymphedema
* Skin lesions at the place where the taping will be applied
* Local sensitivity in the skin sensitivity test to be performed the day before the application
* Chronic kidney failure patients
* Patients with congestive heart failure
* Patients with a body mass index of 30 and above
* Patients who underwent surgery for pathological fractures
* Patients who underwent total knee replacement revision surgery
* Patients who had previously undergone high tibial osteotomy or unicondylar knee replacement surgery
* Patients who underwent surgery due to traumatic arthrosis

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline at 15th, 45th and 90th days in Pain | The clinical evaluation will be made on the 15th, 45th and 90th days
  Visual analogue scale will be used for pain assessment in rest, activity and sleep. The patient will be asked to define the severity of pain in a 10 cm line, from 0 to 10. 0 means no pain and 10 means unbearable pain.
Change from Baseline at 15th, 45th and 90th days in Range of Motion Assessment | The evaluation will be made on the 15th, 45th and 90th days
  range of motion of knee flexion and extension will be measured with digital inclinometer
Change from Baseline at 15th, 45th and 90th days in Edema | The evaluation will be made on the 15th, 45th and 90th days
  edema will be made with measurement of the opposite extremity which will be compared with the tape measure

SECONDARY OUTCOMES:
Change from Baseline at 15th, 45th and 90th days in Complications | The evaluation will be made on the 15th, 45th and 90th days
  Complications such as superficial-deep skin infection or allergic reaction will be evaluated.
Change from Baseline at 15th, 45th and 90th days in Functional Assessment of knee | The evaluation will be made on the 15th, 45th and 90th days
  Functional scores before and after surgery will be assessed with Knee Society Score. The Knee Society Score (KSS) has two components (knee and function scores), each of which is scored separately from 0 to 100, with higher values indicating better outcomes.
Change from Baseline at 15th, 45th and 90th days in Functional Assessment for osteoarthritis. | The evaluation will be made on the 15th, 45th and 90th days
  Functional scores before and after surgery will be assessed with Western Ontario and McMaster Universities Osteoarthritis Index Score. The Western Ontario and McMaster University Osteoarthritis Index (WOMAC) is a disease-specific, self administered, health measure developed to study patients with osteoarthritis in the hip or knee. The domains are pain, stiffness, physical function, social function and emotional function. Every question can be given five alternative answers, which means a total of 0-4 points. The maximum score in the Likert version is 20 points for pain, 8 for stiffness and 68 points for physical function. A maximum score of 100 points occurred when the patient had minimum pain, stiffness and optimal function.
Change from Baseline at 15th, 45th and 90th days in Thermographic measurement | The evaluation will be made on the 15th, 45th and 90th days
  Thermal changes in the skin will be assessed via a thermal camera at the knee region
Change from Baseline at 15th, 45th and 90th days in Inflammatory markers as Interleukin 6 (IL-6) | The evaluation will be made on the 15th, 45th and 90th days
  Inflammatory markers in the blood such as Interleukin 6 (IL-6) will be assessed. The reported values for IL-6 in the blood of healthy people vary between 0 and 43.5 pg/ml.
Change from Baseline at 15th, 45th and 90th days in Inflammatory markers as Sedimentation rate | The evaluation will be made on the 15th, 45th and 90th days
  Inflammatory markers in the blood such as Sedimentation rate, the rate at which they settle is measured as the number of millimeters of clear plasma present at the top of the column after one hour (mm/hr), will be assessed.
Change from Baseline at 15th, 45th and 90th days in Inflammatory markers as C-reactive protein (CRP) | The evaluation will be made on the 15th, 45th and 90th days
  Inflammatory markers in the blood such as C-reactive protein (CRP) will be assessed. CRP concentration is measured in mg/L
Change from Baseline at 15th, 45th and 90th days in Inflammatory markers as Creatine Kinase (CK) | The evaluation will be made on the 15th, 45th and 90th days
  Inflammatory markers in the blood such as Creatine Kinase (CK) will be assessed. Normal range is 22 to 198 U/L (units per liter)

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided